CLINICAL TRIAL: NCT02660359
Title: A Phase III, Multicentre, Randomised, Double Blind, Parallel Group, Placebo Controlled Study To Assess The Efficacy And Safety Of One Or More Intradetrusor Treatments Of 600 Or 800 Units Of Dysport® For The Treatment Of Urinary Incontinence In Subjects With Neurogenic Detrusor Overactivity Due To Spinal Cord Injury Or Multiple Sclerosis
Brief Title: Dysport® Treatment of Urinary Incontinence in Adults Subjects With Neurogenic Detrusor Overactivity (NDO) Due to Spinal Cord Injury or Multiple Sclerosis - Study 2
Acronym: CONTENT2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow recruitment of patients
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D-FR-52120-223; 2015-000507-44 (EudraCT Number)
Record Dates: First submitted 2016-01-14; First posted 2016-01-21 (Estimated); Results first posted 2021-06-16 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Urinary Incontinence; Overactive Bladder
MeSH Terms: conditions — Urinary Incontinence; Urinary Bladder, Overactive | interventions — Botulinum Toxins, Type A; abobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 600 U Dysport® Group (Experimental)
  Interventions: Biological: Botulinum toxin type A
- 600 U Dysport® Placebo Group (Placebo Comparator)
  Interventions: Drug: Placebo
- 800 U Dysport® Group (Experimental)
  Interventions: Biological: Botulinum toxin type A
- 800 U Dysport® Placebo Group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Botulinum toxin type A — 600 U intra detrusor injection in two treatment periods (Initial and Retreatment phase) delivered at 30 injection points.
  Other Names: AbobotulinumtoxinA (Dysport®); Clostridium BTX-A-haemagglutinin complex
  Arms: 600 U Dysport® Group
Biological: Botulinum toxin type A — 800 U intra detrusor injection in two treatment periods (Initial and Retreatment phase) delivered at 30 injection points
  Other Names: AbobotulinumtoxinA (Dysport®); Clostridium BTX-A-haemagglutinin complex
  Arms: 800 U Dysport® Group
Drug: Placebo — AbobotulinumtoxinA Placebo 600 U intra detrusor injection in two treatment periods (Initial and Retreatment phase) delivered at 30 injection points
  Arms: 600 U Dysport® Placebo Group
Drug: Placebo — AbobotulinumtoxinA Placebo 800 U intra detrusor injection in two treatment periods (Initial and Retreatment phase) delivered at 30 injection points
  Arms: 800 U Dysport® Placebo Group

SUMMARY:
The purpose of this study is to provide confirmatory evidence of the safety and efficacy of two Dysport® doses (600 units [U] and 800 U), compared to placebo in reducing urinary incontinence (UI) in adult subjects treated for neurogenic detrusor overactivity (NDO) due to spinal cord injury (SCI) or multiple sclerosis (MS).

ELIGIBILITY:
Key Inclusion Criteria:

* Urinary Incontinence for at least 3 months prior to Screening as a result of Neurogenic Detrusor Overactivity due to Spinal Cord Injury or Multiple Sclerosis.
* Subjects with Spinal Cord Injury must have a stable neurological injury at T1 level or below which occurred at least 6 months prior to Screening.
* Subjects with Multiple Sclerosis must be clinically stable in the investigator's opinion, with no exacerbation (relapse) of MS for at least 3 months prior to Screening.
* Subjects must have had an inadequate response after at least 4 weeks of oral medications used in the treatment of NDO (e.g. anticholinergics, beta-3 agonists) and/or have intolerable side-effects.
* Routinely performing Clean Intermittent Catheterization (CIC) to ensure adequate bladder emptying.
* An average of at least two episodes per day of Urinary Incontinence recorded on the screening bladder diary.

Key Exclusion Criteria:

* Any current condition (other than NDO) that may impact on bladder function.
* Previous or current, tumour or malignancy affecting the spinal column or spinal cord, or any other unstable cause of SCI.
* Any condition that will prevent cystoscopic treatment administration or CIC usage, e.g. urethral strictures.
* Current indwelling bladder catheter, or removal of indwelling bladder catheter less than 4 weeks prior to Screening.
* BTX-A treatment within 9 months prior to Screening for any urological condition (e.g. detrusor or urethral sphincter treatments).
* Any neuromodulation/electrostimulation usage for urinary symptoms/incontinence within 4 weeks prior to Screening. Any implanted neuromodulation device must be switched off at least 4 weeks prior to Screening.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2016-07-08 (Actual); Primary Completion 2018-11-09 (Actual); Study Completion 2019-07-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (82):
- Argentina (5):
  - Instituto Urológico Buenos Aires, Buenos Aires
  - Centro de Urologia, Buenos Aires
  - Centro Urológico Profesor Bengió, Córdoba
  - Hospital Privado - Centro Médico de Córdoba, Córdoba
  - Instituto Médico Rodriguez Alfici, Godoy Cruz
- Australia (2):
  - Prince of Wales Hospital (POWH), Sydney
  - Westmead Hospital, Westmead
- Belgium (3):
  - Antwerp University hospital, Antwerp
  - Hôpital Erasme, Brussels
  - Ourthe-Amblève, Esneux
- Brazil (10):
  - Universidade Estadual de Campinas - Cidade Universitária Zeferino Vaz, Campinas
  - Hospital de Clinicas, Federal University of Paraná, Curitiba
  - Hospital São Vicente de Paulo, Passo Fundo
  - Santa Casa de Misericórdia de Porto Alegre - Hospital Santa Clara, Porto Alegre
  - Hospital Moinhos de Vento, Pôrto Alegre
  - Hospital São Lucas da PUCRS, Pôrto Alegre
  - Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto da Universidade de São Paulo, Ribeirão Preto
  - Faculdade de Medicina do ABC, Santo André
  - Hospital Alemão Oswaldo Cruz, São Paulo
  - Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo
- Chile (3):
  - Clínica Uromed, Santiago
  - Hospital del Trabajador, Santiago
  - Clínica Las Condes, Santiago
- Colombia (5):
  - Solano & Terront Servicios Medicos LTDA- Unidad Integral de Endocrinologia, Bogotá
  - Fundación Valle del Lili, Cali
  - Centro Medico Imbanaco, Cali
  - Asociacion IPS Medicos Internistas de Caldas, Manizales
  - Centro de Investigaciones Clinicas - CIC, Medellín
- France (11):
  - Hôpital Raymond-Poincaré, Garches
  - Centre Hospitalier Régional Universitaire de Lille (CHRU) - Hôpital Claude Huriez, Lille
  - Hôpital de la Conception, Marseille
  - Groupe Hospitalo-Universitaire Pierre Caremau, Nîmes
  - Hopital de la Source, Orléans
  - Hopital Pitie-Salpetriere, Paris
  - Hôpital Tenon, Paris
  - Centre Hospitalier Lyon-Sud, Pierre-Bénite
  - CHU de Rennes - Hôpital Pontchaillou, Rennes
  - CHU de ROUEN - Hôpital Charles Nicolle, Rouen
  - Hôpital Rangueil, Toulouse
- Germany (3):
  - Universitätsklinikum Bonn Klinik und Poliklinik für Urologie, Bonn
  - Kliniken Maria Hilf GmbH - Krankenhaus St. Franziskus, Mönchengladbach
  - Universitätsklinikum Münster, Münster
- Israel (5):
  - Rambam Medical Center, Haifa
  - Carmel Medical Center, Haifa
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center - Davidoff Center, Petah Tikva
  - The Chaim Sheba Medical Center, Ramat Gan
- Lithuania (2):
  - Estetines Chirurgijos Centas, UAB, Kaunas
  - Vilnius University Hospital Santariskiu Klinikos, Vilnius
- Mexico (4):
  - Centro Medico Puerta de Hierro - Colima, Colima
  - Clinstile, S.A. de C.V., Cuauhtémoc
  - Hospital Universitario "Dr. José Eleuterio González", Monterrey
  - Consultorio Privado, Zapopan
- Peru (6):
  - Clínica San Pablo Surco, Lima
  - Clinica Good Hope, Lima
  - Clinica Internacional Sede Lima, Lima
  - Clínica Anglo Americana, Lima
  - Instituto de Ginecología y Reproducción, Lima
  - Unidad de Investigación de la Clínica Internacional Sede San Borja, Lima
- Russia (8):
  - Scientific research institute of urology and interventional radiology n. a. N. A. Lopatkin, Moscow
  - Ministry of healthcare of the Russian Federation, Moscow
  - Penza Regional Clinical Hospital n.a. N.N.Burdenko, Penza
  - Rostov State Medical University, Rostov-on-Don
  - St. Petersburg Research Institute of Phthisiopulmonology, Saint Petersburg
  - Pavlov First Saint Petersburg State Medical University, Saint Petersburg
  - City Hospital No. 40, Saint Petersburg
  - Hospital Orkli, Saint Petersburg
- Spain (7):
  - Complexo Hospitalario Universitario A Coruña, A Coruña
  - Fundacio Puigvert, Barcelona
  - Fundació GAEM, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitari i Politècnic La Fe, Valencia
- Ukraine (2):
  - Municipal Healthcare Institution "Regional Clinical Center of Urology and Nephrology n.a. V.I. Shapoval", Urology Department, Kharkiv
  - Kiev City Clinical Hospital No. 3, Kiev
- United Kingdom (6):
  - NHS Grampian - Aberdeen Royal Infirmary, Aberdeen
  - Bedford Hospital, Bedford
  - National Hospital for Neurology and Neurosurgery - UCL, London
  - Sheffield Teaching Hospitals NHS Foundation Trust - Royal Hallamshire Hospital, Sheffield
  - Royal National Orthopaedic Hospital Trust, Stanmore
  - The Mid Yorkshire Hospitals NHS Trust - Pinderfields Hospital, Wakefield

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized, and study documents will be redacted to protect the privacy of study participants.
  Any requests should be submitted to www.vivli.org for assessment by an independent scientific review board.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and EU or after the primary manuscript describing the results has been accepted for publication, whichever is later.
Access Criteria: Further details on Ipsen's sharing criteria, eligible studies and process for sharing are available here (https://vivli.org/members/ourmembers/).
URL: https://vivli.org/members/ourmembers/

REFERENCES:
- [Derived] Kennelly M, Cruz F, Herschorn S, Abrams P, Onem K, Solomonov VK, Del Rosario Figueroa Coz E, Manu-Marin A, Giannantoni A, Thompson C, Vilain C, Volteau M, Denys P; Dysport CONTENT Program Group. Efficacy and Safety of AbobotulinumtoxinA in Patients with Neurogenic Detrusor Overactivity Incontinence Performing Regular Clean Intermittent Catheterization: Pooled Results from Two Phase 3 Randomized Studies (CONTENT1 and CONTENT2). Eur Urol. 2022 Aug;82(2):223-232. doi: 10.1016/j.eururo.2022.03.010. Epub 2022 Apr 7. PMID 35400537

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 258 subjects with urinary incontinence (UI) caused by neurogenic detrusor overactivity (NDO) due to spinal cord injury (SCI) or multiple sclerosis (MS) were enrolled at 67 study sites worldwide. One of the 258 randomised subjects did not receive any treatment. The study was terminated early by the sponsor due to lack of recruitment.
Pre-assignment Details: Subjects were randomised to 1 of 4 sequences: A) placebo in a double-blind placebo-controlled (DBPC) cycle then Dysport® 600 Units (U) in subsequent double-blind cycles: B) placebo in DBPC cycle then Dysport® 800 U in subsequent cycles: C) Dysport® 600 U in all cycles: D) Dysport® 800 U in all cycles. The minimum retreatment interval was 12 weeks.
Groups:
- Placebo: Subjects were administered placebo on Day 1 of the DBPC cycle. All study treatments were injected into the detrusor muscle via cystoscopy in a total volume of 15 millilitres (mL) divided into 30 injection points of 0.5 mL each. Subjects were followed-up by telephone at Week 1 and Week 4; and attended clinic visits at Week 2, Week 6 (primary study timepoint), and Week 12. Thereafter telephone visits were scheduled every 12 weeks until end of study, or until retreatment was required.
- Dysport® 600 U: Subjects were administered Dysport® 600 U on Day 1 of the DBPC cycle. All study treatments were injected into the detrusor muscle via cystoscopy in a total volume of 15 mL divided into 30 injection points of 0.5 mL each. Subjects were followed-up by telephone at Week 1 and Week 4; and attended clinic visits at Week 2, Week 6 (primary study timepoint), and Week 12. Thereafter telephone visits were scheduled every 12 weeks until end of study, or until retreatment was required.
- Dysport® 800 U: Subjects were administered Dysport® 800 U on Day 1 of the DBPC cycle. All study treatments were injected into the detrusor muscle via cystoscopy in a total volume of 15 mL divided into 30 injection points of 0.5 mL each. Subjects were followed-up by telephone at Week 1 and Week 4; and attended clinic visits at Week 2, Week 6 (primary study timepoint), and Week 12. Thereafter telephone visits were scheduled every 12 weeks until end of study, or until retreatment was required.
Period: Overall Study
Arm/Group | Placebo | Dysport® 600 U | Dysport® 800 U
Started (Subjects randomised and treated in DBPC cycle) | 86 | 86 | 85
Subjects Entered in the Dysport Cycles | 56 | 86 | 85
Completed (Subjects completed the study in the Dysport cycles) | 0 | 0 | 1
Not Completed | 86 | 86 | 84
Not completed — Protocol Deviation | 0 | 0 | 1
Not completed — Sponsor Decision to Terminate Study | 73 | 75 | 71
Not completed — Lack of Efficacy | 1 | 1 | 1
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Other | 2 | 1 | 3
Not completed — Withdrawal by Subject | 7 | 5 | 8
Not completed — Lost to Follow-up | 3 | 3 | 0

BASELINE CHARACTERISTICS:
Population: Modified intention to treat (mITT) population: All randomised subjects who received at least 1 administration of study treatment. Subjects were analysed as randomised (planned treatment).
Groups:
- Placebo: Subjects were administered placebo on Day 1 of the DBPC cycle. All study treatments were injected into the detrusor muscle via cystoscopy in a total volume of 15 mL divided into 30 injection points of 0.5 mL each. Subjects were followed-up by telephone at Week 1 and Week 4; and attended clinic visits at Week 2, Week 6 (primary study timepoint), and Week 12. Thereafter telephone visits were scheduled every 12 weeks until end of study, or until retreatment was required.
- Total: Total of all reporting groups
Arm/Group | Placebo | Dysport® 600 U | Dysport® 800 U | Total
Number analyzed (Participants) | 86 | 86 | 85 | 257
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 80 | 82 | 77 | 239
  >=65 years | 6 | 4 | 8 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.2 (13.16) | 42.5 (12.10) | 42.0 (14.72) | 42.2 (13.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 29 | 30 | 95
  Male | 50 | 57 | 55 | 162
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 8 | 13 | 9 | 30
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 2 | 4 | 4 | 10
  White | 55 | 52 | 56 | 163
  More than one race | 7 | 5 | 3 | 15
  Unknown or Not Reported | 14 | 12 | 12 | 38
Aetiology of NDO [Count of Participants; unit: Participants]
  SCI | 62 | 64 | 65 | 191
  MS | 24 | 22 | 20 | 66

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Weekly Number of UI Episodes at Week 6 of DBPC Cycle
Description: The weekly number of UI episodes was measured using a 7-day bladder diary. Bladder diaries that contained data recorded on at least 5 days were included in the analysis. The least square (LS) mean of the change in weekly number of UI episodes at 6 weeks after the first study treatment was calculated using a mixed model repeated measures (MMRM) analysis.
Time Frame: Baseline and Week 6 of DBPC Cycle
Population: Results are presented for the mITT population (all randomised subjects who received at least 1 administration of study treatment). Subjects were analysed as randomised (planned treatment). Only subjects with data available for analysis at Week 6 of DBPC cycle are presented.
Measure: Least Squares Mean (Standard Error); unit: Weekly UI episodes
Arm/Group | Placebo | Dysport® 600 U | Dysport® 800 U
Number analyzed (Participants) | 76 | 82 | 73
Weekly UI episodes | -12.86 (1.95) | -21.83 (1.91) | -22.62 (1.88)
Statistical Analysis 1: Comparison: Placebo vs Dysport® 600 U; Treatment group, visit (Week 6), treatment-by-visit interaction, recorded stratification factors (aetiology of NDO [SCI or MS], prior intradetrusor [Botulinum toxin [BTX]-naïve or BTX-non-naïve]) and study baseline value (weekly number of UI episodes) as fixed effect variables, and subject as a random effect; Test type: Superiority — If both p-values for the 2 primary tests (the test of Dysport® 800 U vs. placebo and the test of Dysport® 600 U vs. placebo) were lower than 0.05, both were declared statistically significant. If 1 of the primary tests had a p-value greater than or equal to 0.05, then the other test was declared statistically significant if its p-value was lower than 0.025 and only the significant dose continued in the hierarchal testing strategy; p = 0.0001, MMLM; LS Mean Difference = -8.97, 95% CI 2-sided [-13.5 to -4.44]
Statistical Analysis 2: Comparison: Placebo vs Dysport® 800 U; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, MMLM; LS Mean Difference = -9.76, 95% CI 2-sided [-14.41 to -5.12]

2. Secondary Outcome: Percentage of Subjects With No Episodes of UI at Week 6 of DBPC Cycle
Description: The weekly number of UI episodes was measured using a 7-day bladder diary. Bladder diaries that contained data recorded on at least 5 days were included in the analysis. The number of subjects with no UI episodes at 6 weeks after the first study treatment was recorded. Percentage of subjects with no episodes of UI (≥100% Improvement) was calculated as: Total number of subjects with no weekly number of UI episodes at Week 6 / Total number of subjects with any number of UI events at Week 6.
Time Frame: Baseline and Week 6 of DBPC Cycle
Population: as for outcome 1
Measure: Number; unit: Percentage of Subjects
Arm/Group | Placebo | Dysport® 600 U | Dysport® 800 U
Number analyzed (Participants) | 76 | 82 | 73
Percentage of Subjects | 1.3 | 36.6 | 26.0
Statistical Analysis 1: Comparison: Placebo vs Dysport® 600 U; Treatment group, recorded stratification factors, visit, treatment-by-visit interaction, study baseline- by-visit interaction and study baseline weekly number of UI episodes as fixed effect; Test type: Superiority — This secondary endpoint was included in the hierarchical analysis and was tested for both doses at the 0.05 level using a hierarchical methodology; p = 0.0002, Generalised linear mixed model (GLMM); Odds Ratio (OR) = 45.55, 95% CI 2-sided [6.09 to 340.69]
Statistical Analysis 2: Comparison: Placebo vs Dysport® 800 U; Treatment group, recorded stratification factors, visit, treatment-by-visit interaction, study baseline-by-visit interaction and study baseline weekly number of UI episodes as fixed effect; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.0009, GLMM; Odds Ratio (OR) = 31.69, 95% CI 2-sided [4.17 to 240.58]

3. Secondary Outcome: Percentage of Subjects With a UI Response at Improvement Levels ≥30%, ≥50%, and ≥75% at Week 6 of the DBPC Cycle
Description: The weekly number of UI episodes was measured using a 7-day bladder diary. Bladder diaries that contained data recorded on at least 5 days were included in the analysis. The percentage of subjects showing an improvement of ≥30%, ≥50% and ≥75% was calculated as: Total number of subjects with UI response level >=30% or >=50% or >=75% improvement at Week 6 / Total number of subjects with any UI response at Week 6.
Time Frame: Baseline and Week 6 of DBPC Cycle
Population: as for outcome 1
Measure: Number; unit: Percentage of Subjects
Arm/Group | Placebo | Dysport® 600 U | Dysport® 800 U
Number analyzed (Participants) | 76 | 82 | 73
Percentage of Subjects
  ≥30% Improvement | 55.3 | 81.7 | 76.7
  ≥50% Improvement | 38.2 | 72.0 | 61.6
  ≥75% Improvement | 17.1 | 62.2 | 50.7
Statistical Analysis 1: Comparison: Placebo vs Dysport® 600 U; Treatment comparison at ≥30% Improvement Level: Dysport® 600 U versus Placebo; Test type: Superiority — Treatment group, recorded stratification factors, visit, treatment-by-visit interaction, study baseline-by-visit interaction and study baseline weekly number of UI episodes as fixed effect; p = 0.0007, GLMM — This secondary endpoint was not included within the hierarchical testing procedure and was analysed for exploratory purposes only to compare each Dysport® dose to placebo at a 0.05 type one error rate; Odds Ratio (OR) = 3.55, 95% CI 2-sided [1.72 to 7.34]
Statistical Analysis 2: Comparison: Placebo vs Dysport® 800 U; Treatment comparison at ≥30% Improvement Level: Dysport® 800 U versus Placebo; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.0037, GLMM — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 2.94, 95% CI 2-sided [1.43 to 6.07]
Statistical Analysis 3: Comparison: Placebo vs Dysport® 600 U; Treatment comparison at ≥50% Improvement level: Dysport® 600 U versus Placebo; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p < 0.0001, GLMM — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 3.98, 95% CI 2-sided [2.03 to 7.79]
Statistical Analysis 4: Comparison: Placebo vs Dysport® 800 U; Treatment comparison at ≥50% Improvement level: Dysport® 800 U versus Placebo; Test type: Superiority — Treatment group, recorded stratification factors, visit, treatment-by- visit interaction, study baseline-by-visit interaction and study baseline weekly number of UI episodes as fixed effect; p = 0.0034, GLMM — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 2.73, 95% CI 2-sided [1.40 to 5.33]
Statistical Analysis 5: Comparison: Placebo vs Dysport® 600 U; Treatment comparison at ≥75% Improvement level: Dysport® 600 U versus Placebo; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p < 0.0001, GLMM — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 7.38, 95% CI 2-sided [3.5 to 15.58]
Statistical Analysis 6: Comparison: Placebo vs Dysport® 800 U; Treatment comparison at ≥75% Improvement level: Dysport® 800 U versus Placebo; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p < 0.0001, GLMM — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 5.28, 95% CI 2-sided [2.48 to 11.24]

4. Secondary Outcome: Median Time Between Treatments
Description: Duration of effect for time between treatments was calculated by: (the date of the first retreatment visit - date of first treatment administration in the DBPC cycle). The median number of days between treatments was determined and subjects with no retreatment were censored at the last visit.
Time Frame: Day of first treatment (baseline) to day of retreatment, up to 2 years
Population: Results are presented for the mITT population (all randomised subjects who received at least 1 administration of study treatment). Subjects were analysed as randomised (planned treatment).
Measure: Median (Full Range); unit: Days
Arm/Group | Placebo | Dysport® 600 U | Dysport® 800 U
Number analyzed (Participants) | 86 | 86 | 85
Days | 132.0 [8.0 to 644.0] | 238.5 [57.0 to 651.0] | 210.0 [56.0 to 649.0]

5. Secondary Outcome: Mean Change From Baseline in Volume Per Void at Week 6 of DBPC Cycle
Description: The volume per void was measured during one 24-hour period of the 7-day bladder diary. The LS mean of the change in volume per void at 6 weeks after the first study treatment was calculated using a MMRM analysis.
Time Frame: Baseline and Week 6 of DBPC Cycle
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Placebo | Dysport® 600 U | Dysport® 800 U
Number analyzed (Participants) | 74 | 77 | 72
mL | -6.00 (17.80) | 90.14 (17.45) | 84.78 (17.22)
Statistical Analysis 1: Comparison: Placebo vs Dysport® 600 U; Treatment group, visit (Week 6), treatment-by-visit interaction, recorded stratification factors (aetiology of NDO [SCI or MS], prior intradetrusor [BTX-naïve or BTX-non-naïve]) and study baseline value (total volume per void) as fixed effect variables, and subject as a random effect; Test type: Superiority — This secondary endpoint was not included within the hierarchical testing procedure and was analysed for exploratory purposes only to compare each Dysport® dose to placebo at a 0.05 type one error rate; p < 0.0001, MMRM; LS Mean Difference = 96.14, 95% CI 2-sided [53.10 to 139.19]
Statistical Analysis 2: Comparison: Placebo vs Dysport® 800 U; [analysis description as in outcome 5, analysis 1]; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p < 0.0001, MMRM; LS Mean Difference = 90.78, 95% CI 2-sided [47.07 to 134.48]

6. Secondary Outcome: Mean Change From Baseline in Maximum Cystometric Capacity (MCC) at Week 6 of DBPC Cycle
Description: Subjects included in the urodynamic subset (84.9% of randomised subjects) had a standardised urodynamic filling cystometry assessment at baseline (Screening) and again at Week 6 to determine the MCC. The LS mean of the change in MCC at 6 weeks after the first study treatment was calculated using an analysis of covariance (ANCOVA).
Time Frame: Baseline and Week 6 of DBPC Cycle
Population: Results are presented for the urodynamic population (all subjects in the mITT population included in the urodynamic subset at randomisation). Subjects were analysed as randomised (planned treatment). Only subjects with data available for analysis at Week 6 of DBPC cycle are presented.
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Placebo | Dysport® 600 U | Dysport® 800 U
Number analyzed (Participants) | 62 | 76 | 63
mL | 3.5 (22.83) | 178.5 (21.38) | 171.9 (21.58)
Statistical Analysis 1: Comparison: Placebo vs Dysport® 600 U; Treatment group, recorded stratification factors (aetiology of NDO [SCI or MS], prior intradetrusor [BTX- naïve or BTX-non-naïve]) and baseline value of MCC as covariates; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p < 0.0001, ANCOVA; LS Mean Difference = 175.0, 95% CI 2-sided [122.90 to 227.0]
Statistical Analysis 2: Comparison: Placebo vs Dysport® 800 U; [analysis description as in outcome 6, analysis 1]; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p < 0.0001, ANCOVA; LS Mean Difference = 168.4, 95% CI 2-sided [113.6 to 223.1]

7. Secondary Outcome: Mean Change From Baseline in Maximum Detrusor Pressure (MDP) During Storage at Week 6 of DBPC Cycle
Description: Subjects included in the urodynamic subset (84.9% of randomised subjects) had a standardised urodynamic filling cystometry assessment at baseline (Screening) and again at Week 6 to determine the MDP. The LS mean of the change in MDP at 6 weeks after the first study treatment was calculated using an ANCOVA.
Time Frame: Baseline and Week 6 of DBPC Cycle
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: centimetres of water
Arm/Group | Placebo | Dysport® 600 U | Dysport® 800 U
Number analyzed (Participants) | 54 | 71 | 57
centimetres of water | -3.7 (3.84) | -36.7 (3.48) | -36.2 (3.51)
Statistical Analysis 1: Comparison: Placebo vs Dysport® 600 U; Treatment group, recorded stratification factors (aetiology of NDO [SCI or MS], prior intradetrusor [BTX- naïve or BTX-non-naïve]) and baseline value of MDP as covariates; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p < 0.0001, ANCOVA; LS Mean Difference = -32.9, 95% CI 2-sided [-41.5 to -24.4]
Statistical Analysis 2: Comparison: Placebo vs Dysport® 800 U; [analysis description as in outcome 7, analysis 1]; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p < 0.0001, ANCOVA; LS Mean Difference = -32.5, 95% CI 2-sided [-41.5 to -23.4]

8. Secondary Outcome: Mean Change From Baseline in Volume at First Involuntary Detrusor Contraction (Vol@1stIDC) at Week 6 of DBPC Cycle
Description: Subjects included in the urodynamic subset (84.9% of randomised subjects) had a standardised urodynamic filling cystometry assessment at baseline (Screening) and again at Week 6 to determine the Vol@1stIDC which is the instilled volume when first IDC commences. Subjects who did not exhibit a post-treatment IDC at Week 6 had Vol@1stIDC imputed using the recorded corrected MCC volume at Week 6. The LS mean of the change in Vol@1stIDC at 6 weeks after the first study treatment was calculated using an ANCOVA.
Time Frame: Baseline and Week 6 of DBPC Cycle
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Placebo | Dysport® 600 U | Dysport® 800 U
Number analyzed (Participants) | 60 | 72 | 58
mL | 15.9 (23.34) | 168.7 (22.09) | 185.5 (22.80)
Statistical Analysis 1: Comparison: Placebo vs Dysport® 600 U; Treatment group, recorded stratification factors (aetiology of NDO [SCI or MS], prior intradetrusor [BTX- naïve or BTX-non-naïve]) and baseline value of Vol@1stIDC as covariates; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p < 0.0001, ANCOVA; LS Mean Difference = 152.8, 95% CI 2-sided [99.2 to 206.5]
Statistical Analysis 2: Comparison: Placebo vs Dysport® 800 U; [analysis description as in outcome 8, analysis 1]; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p < 0.0001, ANCOVA; LS Mean Difference = 169.7, 95% CI 2-sided [111.7 to 227.6]

9. Secondary Outcome: Percentage of Subjects With No Involuntary Detrusor Contraction (IDCs) During Storage at Week 6 of DBPC Cycle
Description: Subjects included in the urodynamic subset (84.9% of randomised subjects) had a standardised urodynamic filling cystometry assessment at baseline (Screening) and again at Week 6 to determine the occurrence of IDCs. The percentage of subjects without IDCs at 6 weeks after the first study treatment was recorded.
Time Frame: Baseline and Week 6 of DBPC Cycle
Population: as for outcome 6
Measure: Number; unit: Percentage of Subjects
Arm/Group | Placebo | Dysport® 600 U | Dysport® 800 U
Number analyzed (Participants) | 59 | 74 | 58
Percentage of Subjects | 3.4 | 52.7 | 50.0
Statistical Analysis 1: Comparison: Placebo vs Dysport® 800 U; [analysis description as in outcome 2, analysis 2]; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p < 0.0001, GLMM; Odds Ratio (OR) = 31.1, 95% CI 2-sided [7.05 to 137.09]
Statistical Analysis 2: Comparison: Placebo vs Dysport® 800 U; Treatment group, recorded stratification factors, visit, treatment-by-visit interaction, study baseline-by- visit interaction and study baseline weekly number of UI episodes as fixed effect; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p < 0.0001, GLMM; Odds Ratio (OR) = 28.08, 95% CI 2-sided [6.24 to 126.25]

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events are presented for the full DBPC cycle (i.e. approximately 32 weeks for both Dysport® groups and approximately 19 weeks for the Placebo group).
Description: The safety population included all subjects who received at least 1 administration of study treatment (including only partial administration). Safety subjects were analysed according to their actual treatment received. One subject randomised to placebo received Dysport 600 U, and 1 subject randomised to Dysport 800 U did not receive treatment and was not included in the safety population. Number of deaths (all causes) is presented for the duration of the study (up to a maximum of 115 weeks).
Arm/Group | Placebo | Dysport® 600 U | Dysport® 800 U
All-Cause Mortality (participants affected / at risk) | 0/85 | 1/87 | 0/85
Serious Adverse Events (participants affected / at risk) | 0/85 | 9/87 | 8/85
Other Adverse Events (participants affected / at risk) | 34/85 | 40/87 | 42/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=85) | Dysport® 600 U (N=87) | Dysport® 800 U (N=85)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Multiple sclerosis relapse (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Multiple sclerosis (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (2) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis chronic (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Perineal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Testicular abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Orchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=85) | Dysport® 600 U (N=87) | Dysport® 800 U (N=85)
Haemorrhage (Vascular disorders) | 0 (0) | 2 (2) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 2 (2) | 1 (1)
Anaesthetic complication cardiac (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1)
Nitrite urine present (Investigations) | 2 (2) | 2 (2) | 0 (0)
Blood urine present (Investigations) | 2 (2) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 3 (5)
Muscle spasticity (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 3 (5) | 2 (2)
Fatigue (General disorders) | 0 (0) | 1 (1) | 2 (2)
Malaise (General disorders) | 1 (1) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 3 (7) | 4 (4)
Constipation (Gastrointestinal disorders) | 1 (1) | 4 (4) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (2) | 2 (2)
Abdominal pain lower (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2)
Haematuria (Renal and urinary disorders) | 4 (4) | 5 (5) | 4 (4)
Leukocyturia (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (5) | 5 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 17 (21) | 19 (24) | 22 (34)
Bacteriuria (Infections and infestations) | 0 (0) | 6 (6) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 4 (4)
Influenza (Infections and infestations) | 5 (5) | 2 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Pharyngitis (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Bladder pain (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This study was terminated early by the sponsor on 04 October 2018, due to slow subject recruitment (258 subjects randomised compared to 330 planned subjects). Only primary and key secondary efficacy analyses were performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-04-16): https://cdn.clinicaltrials.gov/large-docs/59/NCT02660359/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-21): https://cdn.clinicaltrials.gov/large-docs/59/NCT02660359/SAP_001.pdf